CLINICAL TRIAL: NCT04979273
Title: The Role of Hypertonic Dextrose Spray as Endoscopic Topical Hemostatic Agent for Acute Non-Variceal Upper Gastrointestinal Bleeding: A Randomized Controlled Trial
Brief Title: The Role of Hypertonic Dextrose Spray as Endoscopic Topical Hemostatic Agent for Acute Non-Variceal Upper GI Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Hasan Maulahela, MD, Head of Gastrointestinal Endoscopy Center FKUI-RSCM, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-02-0130
Record Dates: First submitted 2021-07-02; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Gastro Intestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Glucose; Water; Epinephrine; Solutions; Injections; Argon Plasma Coagulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients within control group will be given adrenaline 1:20.000 injection, followed by thermocoagulation or hemoclip
  Interventions: Drug: Adrenaline 1 Mg/mL Solution for Injection; Procedure: argon plasma coagulation; Procedure: Hemoclip
- Dextrose group (Experimental): Patients within this group will be given adrenaline 1:20.000 injection, followed by dextrose 40% spray
  Interventions: Drug: Dextrose 40 % in Water; Drug: Adrenaline 1 Mg/mL Solution for Injection

INTERVENTIONS:
Drug: Dextrose 40 % in Water — injection of adrenaline 1:20.000, followed by dextrose 40% spray
  Arms: Dextrose group
Drug: Adrenaline 1 Mg/mL Solution for Injection — injection of adrenaline 1:20.000, followed by thermocoagulation or hemoclip
Procedure: argon plasma coagulation — Thermocoagulation
  Arms: Control Group
Procedure: Hemoclip — Hemoclip
  Arms: Control Group

SUMMARY:
This study is conducted to evaluate the effectivity of hypertonic dextrose spray as an endoscopic topical hemostatic agent, compared to conventional agent (adrenaline injection, followed by hemoclip or thermocoagulation), in patients with acute non-variceal upper GI bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute non-variceal upper gastrointestinal bleeding caused by peptic or duodenal ulcer, polyps, tumors or malignancy
* Patients consented to study participation

Exclusion Criteria:

* Patients with thrombocytopenia (thrombocyte count <100.000 cells/ul) and other forms of coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Hemostatic success | 5 minute
  Number of participants whose bleeding stops within five minutes after intervention is given. Outcome is assessed by independent assessor (not the endoscopy operator), who also attend the endoscopy session and could observe whether the bleeding stops.

SECONDARY OUTCOMES:
Re-bleeding | 7 days
  Number of participants who experience decrease in hemoglobin >1g/dl or need additional hemostatic endoscopy within one week after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Maulahela, MD, Principal Investigator — Dr Cipto Mangunkusumo General Hospital
Locations (1):
- Dr. Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided